CLINICAL TRIAL: NCT02006004
Title: Epidemiologic Registry of Patients Diagnosed With Acute Myeloid Leukemia (PETHEMA LMA 2013)
Brief Title: Epidemiologic Registry PETHEMA LMA 2013
Status: Completed | Type: Observational
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: PETHEMA LMA 2013
Record Dates: First submitted 2013-11-26; First posted 2013-12-09 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: AML
Keywords: AML

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Epidemiologic and retrospective multicenter registry of all patients diagnosed with de novo or secondary AML in the PETHEMA Group institutions. This study is a non-interventional research regarding diagnosis and therapeutic approach

DETAILED DESCRIPTION:
To perform this registry, every patient diagnosed with AML in the participant institutions, regardless type of AML and treatment administered, must be reported. It will be required to registry the main characteristics of the patients and AML at diagnosis, as cytomorphologic, immunophenotypic, and cytogenetic results, according to the habitual practice of the centers. The treatment which has been administered by every center of the PETHEMA Group, even when it is considered as supportive care, and evolution of the disease will also be reported (relapse o death). PETHEMA Group will input all the reported information in data bases with the appropriate security.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with acute myeloid leukemia

Exclusion Criteria:

no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2012-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Characteristics of the patients diagnosed with AML | 3 years
  To realize an epidemiologic and retrospective study to assess the characteristics of the patients diagnosed with AML and their disease, regardless the age or treatment

SECONDARY OUTCOMES:
Prognosis factors | 3 years
  To correlate clinical and biological features with outcome and evolution of the patients.
Risk factors | 3 years
  To identify and confirm the risk factors which are involved in the evolution of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sanz Miguel Angel, DR, Principal Investigator — Hospital La Fe
Locations (1):
- Hospital La Fe, Valencia, Valencia, Spain